CLINICAL TRIAL: NCT05212012
Title: A Phase I/II Trial of D,L-MEthadone and mFOLFOX6 in Treatment of Advanced Colorectal Cancer - The AIO-MEFOX Trial (AIO-KRK-0119)
Brief Title: D,L-MEthadone and mFOLFOX6 in Treatment of Advanced Colorectal Cancer
Acronym: MEFOX
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-KRK-0119; 2024-519509-37-00 (EU CTIS Number)
Record Dates: First submitted 2021-11-02; First posted 2022-01-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Chemo-refractory Colorectal Carcinoma
Keywords: chemo-refractory; colorectal carcinoma; D,L-methadone; mFOLFOX6
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Maximum Tolerated Dose

STUDY DESIGN:
Intervention Model Description: Phase I: 3+3 dose escalation study (non-randomized) - max. 18 participant
  after Phase I start with a Amendment Phase II: Open-label, 2:1 randomized, controlled trial - 64 participant Patients in the mFOLFOX6 alone arm are allowed to cross over and receive methadone hydrochloride in combination with mFOLFOX6 upon disease progress
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D,L-methadonehydrochloride + mFOLFOX6 (Experimental): Dose Level D,L-methadone hydrochloride (Methasan® 10 mg/ml) In dose level I a maximum of 30 mg/day (15 mg (1,5 ml) 1-0-1) In dose level II a maximum of 35 mg/ day (17.5 mg (1,75 ml) 1-0-1) In dose level III a maximum of 40 mg/day (20 mg (2,0 ml) 1-0-1)
  Treatment with mFOLFOX6 every two weeks; will be administered:
  Oxaliplatin at a dose of 85 mg/m² iv over two hours (day 1) LV at a dose of 400 mg/m² iv over two hours (day 1) 5-FU at a dose of 2400 mg/m² iv over 46 hours (day 1-3)
  Interventions: Drug: Maximum tolerated dose, MTD: D,L-methadone hydrochloride (Methasan® 10 mg/ml)

INTERVENTIONS:
Drug: Maximum tolerated dose, MTD: D,L-methadone hydrochloride (Methasan® 10 mg/ml) — Dose Level D,L-methadone hydrochloride (Methasan® 10 mg/ml) In dose level I a maximum of 30 mg/day (15 mg (1,5 ml) 1-0-1) In dose level II a maximum of 35 mg/ day (17.5 mg (1,75 ml) 1-0-1) In dose level III a maximum of 40 mg/day (20 mg (2,0 ml) 1-0-1)

SUMMARY:
This is a phase I/II-trial with D,L-methadone and mFOLFOX6 in the treatment of patients with histologically confirmed chemo-refractory colorectal carcinoma.

The aim of the phase-I trial is to evaluate the toxicity-profile and the dose-limiting toxicity of D,L-methadone combined with mFOLFOX6. Furthermore, to estimate the maximum tolerated dose and the recommended dose for phase-II-trial in the treatment of patients with histologically confirmed colorectal carcinoma not amenable to or progressing while having received all standard therapies.

The primary endpoint of the randomized phase-II study is to determine the disease control rate 12 weeks after randomization of patients with histologically confirmed advanced colorectal carcinoma upon treatment with D,L methadone plus mFOLFOX6 versus mFOLFOX6 alone. Overall response rate according to RECIST1.1, progression free survival (PFS), overall survival (OS), quality of life (QoL) according to the EORTC QLQc30 questionnaire, patient-reported outcomes and safety will be evaluated as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, histologically confirmed, metastatic colorectal carcinoma not suitable for resection and chemorefractory or Previously employed chemotherapy regimens and agents should comprise the following: Fluoropyrimidines, oxaliplatin, irinotecan, antiangiogenic agents (bevacizumab, aflibercept or ramucirumab), anti-EFGR-mAbs (in case of all-Ras-wildtype and left-sided primary tumor) and Trifluridin/Tipiracil (TAS102)
* Microsatellite stable subset (MSS) of colorectal cancer
* Prior antineoplastic therapy or radiochemotherapy is allowed up to two weeks prior to start of the study medication. However, for the phase II part of the trial, failure of this strategy must be confirmed. In case of prior radiotherapy/radiochemotherapy the target lesion used for tumor evaluation must not be in the radiation field.
* There must be an oxaliplatin free period of at least 6 months prior to start of the study medication.
* No polyneuropathy of > grade 1
* Tumor-related ECOG performance status 0-2
* Anticipated life expectancy ≥ 12 weeks
* Creatinine clearance ≥ 30 ml/min
* Serum total bilirubin level ≤ 3 x ULN.
* ALT and AST ≤ 2.5 x ULN or ≤ 5.0 x ULN in the presence of liver metastasis (established after adequate biliary drainage)
* White blood cell count ≥ 3.5 x 106/ml, neutrophil granulocytes count ≥ 1,5 x 106/ml, platelet count ≥ 100 x 106/ml
* Pain that has to be controllable without concomitant use of opioids
* Signed informed consent according to ICH/GCP and national/local regulations (participation in translational research is obligate)
* None of the following concomitant medications: MAO-B-Inhibitors, strong inductors or inhibitors of CYP3A4, antiarrhythmic drugs of class I and III or other drugs that have potential for QT-prolongation
* Age ≥ 18 years
* At least one measurable target lesion according to RECIST 1.1. Pre-irradiated or locally treated lesions must not be used as target lesions.

Exclusion Criteria:

* Microsatellite unstable CRC (MSIhigh)
* Chronic infectious diseases, immune deficiency syndromes
* Polyneuropathy >grade I according to CTCAE V4.03
* Premalignant hematologic disorders, e.g. myelodysplastic syndrome
* Disability to understand and sign written informed consent document
* Past or current history of malignancies except for the indication under this study and curatively treated:

  * Basal and squamous cell carcinoma of the skin
  * In-situ carcinoma of the cervix
  * Other malignant disease without recurrence after at least 3 years of follow-up
* Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) 6 months before enrollment
* History of or evidence upon physical examination of CNS disease unless adequately treated (e.g. primary brain tumor, seizure not controlled with standard medical therapy or history of stroke).
* Severe non-healing wounds, ulcers or bone fractions
* Evidence of bleeding diathesis or coagulopathy
* Patients not receiving therapeutic anticoagulation must have an INR ≤ 1.4 or PTT ≤ 40 sec within 28 days prior to randomization. The use of full dose anticoagulants is allowed as long as the INR or PTT is within therapeutic limits (according to the medical standard in the institution)
* Major surgical procedures or significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgical procedure during the course of the study.
* Pregnancy or breastfeeding women.
* Use of cannabinoids because of overlapping and /or potentiating of potential side effects
* Concomitant daily use of opioids in the last 3 months including methadone prior start of study medication
* Subjects with known allergies to the study drugs or to any of its excipients.
* Treatment with another investigational drug or participation in another interventional trial (within the 14 days prior randomization or 5 plasma half-lifes of the used investigational drug, whatever is longer)
* Congenital QT-syndrome.
* Alcohol abuse.
* Bronchial asthma.
* Liver cirrhosis > Child-Pugh classification A.
* Any psychological, familial, sociological or geographical condition potentially compromising compliance with the study protocol and the follow-up schedule; those conditions should be discussed with the patient prior to registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the recommended dose for phase-II-trial | 18 months
  Evaluation of the toxicity-profile of D,L-methadone and the dose-limiting toxicity (DLT) in combination with mFOLFOX6
Disease control rate 12 weeks after randomization (ITT-population) | 12 weeks after randomization
  Evaluation of the disease control rate of D,L-methadone plus mFOLFOX6 compared to mFOLFOX6 alone in the treatment of patients with advanced colorectal cancer. The disease control rate is defined as response (CR or PR) or stabilization (SD) of the tumor disease at 12 weeks after randomization (DCR) according to RECIST1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) 12 weeks after randomization (per-protocol-population) | 12 weeks
  The disease control rate is defined as response (CR or PR) or stabilization (SD) of the tumor disease at 12 weeks after randomization (DCR) according to RECIST1.1
Overall response rate | 46 months
  All tumor evaluation is performed according to RECIST 1.1
patient diary | 46 months
  Collection compliance with a diary
Progression-free survival | after 46 months
  Progression-free survival (PFS) will be defined as the time from randomization to the time of progress (according to RECIST 1.1) or death, or to the date of last tumor assessment without any such event (censored observation)
Overall survival | 46 months
  The duration of overall survival (OS) will be determined by measuring the time interval from randomization to the date of death or last observation (censored)
Quality of life assessment | 46 months
  EORTC QLQ-C30 ("European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30)" ).
  The EORTC QLQ-C30 is composed of a global health status/QoL-score, five function scales, three symptom scales and five single items (dyspnea, insomnia, appetite loss, constipation, diarrhea). Each item has four response alternatives: (1) "not at all", (2) "a little", (3) "quite a bit", and (4) "very much" - except the two items of the global health-status/quality of life scale which have response options ranging from (1) "very poor" to (7) "excellent".
Adverse events | 46 months
  Evaluation of the safety- and tolerability profile

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Seufferlein, Prof.Dr.med., Principal Investigator — Ulm University Hospital, Department of Internal Medicine I
Locations (3):
- Germany (3):
  - Universitätsklinikum Hamburg Eppendorf - II. Med., Hamburg
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Universitätsklinikum Ulm - Innere Med. I, Ulm

IPD SHARING:
Plan to Share IPD: No